CLINICAL TRIAL: NCT04903483
Title: Anesthesia of Endolaryngeal Laser Surgery and Perioperative Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Timea Bocskai, senior lecturer, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 6218-2021
Record Dates: First submitted 2021-05-22; First posted 2021-05-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia
Keywords: laser, anesthesia, bispectral index, postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: the side effects of endolaryngeal laser surgery's anesthesia with or without bispectral index monitoring in patients with smoking
Who Masked: Participant
Masking Description: anesthesia with target-controlled infusion (propofol) with or without the depth of anesthesia (bispectral index) monitoring and evaluation of vital parameters, side effects, and postoperative delirium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- target-controlled infusion (propofol) with depth of anesthesia monitoring (Other): In this group, propofol dosing is adjusted with bispectral index monitoring.
  Interventions: Other: bispectral index monitoring
- target-controlled infusion (propofol) without depth of anesthesia monitoring (Other): In this group, propofol dosing is adjusted without bispectral index monitoring.
  Interventions: Other: bispectral index monitoring

INTERVENTIONS:
Other: bispectral index monitoring — intraoperative single-channel electroencephalography monitoring of the depth of anesthesia
  Other Names: depth of anesthesia

SUMMARY:
Investigators analyze the anesthesia of the endolaryngeal laser surgery in patients with smoking with or without monitoring of depth of anesthesia (bispectral index)

DETAILED DESCRIPTION:
All participants are informed about the investigation and are signed the Informed Consent before anesthesia. The study takes place at the Department of Otorhinolaryngology, University of Pecs, Hungary. Between June 2021 and May 2022 ASA I or II patients aged 18-65 years, scheduled for elective endolaryngeal laser surgery with TCI (target-controlled infusion, propofol). Exclusion criteria are epilepsy, psychiatric illness, cerebrovascular or congenital neuromuscular disease. Participants are randomized to two anesthetic groups, anesthesia with or without bispectral index monitoring.

ELIGIBILITY:
Inclusion Criteria:

* endolaryngeal laser surgery with target-controlled anesthesia

Exclusion Criteria:

* epilepsy, psychiatric illness, cerebrovascular or congenital neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
circulation | through study completion, an average of 1 year
  blood pressure (mmHg)
cardiac function | through study completion, an average of 1 year
  pulse rate (beats/minute)
oxygenization | through study completion, an average of 1 year
  oxygen saturation (%)
ventilation | through study completion, an average of 1 year
  end-tidal carbon-dioxide (mmHg)
depth of anesthesia | through study completion, an average of 1 year
  bispectral index level (number between 1-100), the target intraoperative level 40-60, lower and higher are worse

SECONDARY OUTCOMES:
cognitive functions | through study completion, an average of 1 year
  cognitive functions test (Montreal Cognitive Assessment) score (number between 0-30, minimum=0, maximum=30), higher number is better

CONTACTS AND LOCATIONS:
Overall Officials: Burian Andras, MD, Study Chair — University of Pecs Department of ENT
Locations (2):
- Hungary (2):
  - Department of Anaesthesiology and Intensive Therapy, Pécs, Ifjuság Str.13.
  - PTE Department of ENT, Pécs